CLINICAL TRIAL: NCT00870714
Title: Neoadjuvant Therapy With Docetaxel and Ketoconazole in Patients With High-Risk Prostate Cancer: A Pilot Study
Acronym: IST 16167
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kansas City Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Sanofi (Industry)
Responsible Party: Peter VanVeldhuizen, M.D./Principal Investigator, Kansas City VAMC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sanofi-Aventis IST 16167
Record Dates: First submitted 2008-07-24; First posted 2009-03-27 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Eligible patients with high-risk prostate cancer who are scheduled to undergo radical prostatectomy will receive four cycles of therapy with ketoconazole and docetaxel prior to surgery resection
  Interventions: Drug: Docetaxel; Drug: Ketoconazole

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 55mg/m2 to be given IV as a one-hour infusion to be repeated every 21 days for four treatment cycles.
Drug: Ketoconazole — Ketoconazole 400mg P.O. BID daily to start on day 2 following the first docetaxel treatment. In patients who experience no grade 2 or higher toxicity, the ketoconazole dose will be increased to 400mg TID on day 2 following cycle #2 of docetaxel. This will be continued daily until completion of study treatment.

SUMMARY:
Eligible patients with high-risk prostate cancer who are scheduled to undergo radical prostatectomy will receive four cycles of therapy with ketoconazole and docetaxel prior to surgery resection. A cycle of therapy is defined as 21 days (three weeks). Pharmacokinetic analysis will be performed with the first and second cycle of therapy. All patients will be evaluated for toxicity, tumor response, and recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven adenocarcinoma of the prostate.
* Patients must meet at least one of the following high risk criteria:

  * PSA > 20
  * Gleason score 8 or greater
  * Presence of pathological Gleason grade 4 or higher as the majority sum on biopsy core
  * Greater than 50% of cores at time of biopsy positive for cancer
  * Clinical Stage T3 Disease
  * Patients must have PS of 0-1(ECOG) and medically deemed a surgical candidate for radical prostatectomy.
  * Age > or = to 18.
  * Patients with a pre-existing peripheral neuropathy of equal to or greater than grade two are ineligible.
  * Serum Creatinine must be < or equal to 2.0mg/dl.
  * Patients must currently not receiving any drug which is metabolized by cytochrome P450-3A4 including the statins, cyclosporin, terfenadine and erythromycin.
  * Prior to receiving any dose of docetaxel, patients should have absolute neutrophil counts > 1,500, hemoglobin > 8.0 g/dl and platelet counts > 100,000/mm3.
  * Patients with bilirubin elevated above institutional upper limit of normal (ULN)must be excluded. Transaminases (SGOT and/or SGPT) may be up to 5.0 x institutional upper limit of normal (ULN) if alkaline phosphatase is < ULN, or alkaline phosphatase may be up to 5 x ULN if transaminases are < ULN. However, patients who have both transaminase elevation > 1.5 x ULN and alkaline phosphatase > 2.5 x ULN are not eligible for this study (due to decrease clearance of docetaxel and increased risk of toxicity).
  * Patients receiving concurrent warfarin are eligible but require monitoring of protime on a weekly basis.
  * Patients with clinical stage T4 disease are not eligible.
  * Patients must not had have received prior treatment with surgery, radiation or hormone deprivation.
  * Patients with other primary malignancies previously treated with chemotherapeutic agents are not eligible.
  * Patients must not have had a history of peptic ulcer disease requiring treatment with surgery or endoscleral.
  * Patients requiring corticosteroids for other systemic diseases are not eligible.
  * Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 are not eligible.
  * All patients must sign informed consent.
  * Men of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-09; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
To determine the pathologic response rate of neoadjuvant therapy with the combination of docetaxel and ketoconazole given to patients who are at a high risk of recurrence of prostate cancer. | One year

SECONDARY OUTCOMES:
To assess in preliminary fashion whether of this treatment will decrease the incidence of biochemical recurrence and provide a survival benefit as compared to patients with local treatment only or other adjuvant therapies. | One Year

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas City VAMC, Kansas City, Missouri, United States